CLINICAL TRIAL: NCT00623818
Title: fMRI Investigation of Cortical Reorganization and Phantom Limb Pain Following Amputation
Brief Title: Mirror Therapy for Phantom Limb Pain
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080052; 08-M-0052
Record Dates: First submitted 2008-02-24; First posted 2008-02-26 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12-10

CONDITIONS: Amputation
Keywords: Mirror Therapy; Phantom Limb Pain; Amputee; Healthy Volunteer; HV
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study, conducted at the National Institutes of Health (NIH) and at Walter Reed Army Medical Center (WRAMC), will explore the phenomenon of phantom limb pain (a continued feeling of pain in an amputated limb) and will use functional magnetic resonance imaging (fMRI) to investigate the effect of mirror therapy on phantom limb pain.

Right-handed people between 18 and 75 years of age who are in the WRAMC Military Amputee Research Program and healthy control subjects may be eligible for this study. Participants undergo the following procedures:

Amputees

* Questionnaires to assess strength of handedness and footedness and pain perception.
* Mirror therapy for phantom limb pain five times a week for 4 weeks in 15-minute sessions.
* MRI and fMRI scans before starting mirror therapy, after 2 weeks of therapy and after 4 weeks of therapy. MRI uses a magnetic field and radio waves to image brain tissue. The subject lies on a table that can slide in and out of the scanner (a metal cylinder). The structural MRI scan lasts about 30 minutes. For fMRI, the subject performs tasks while in the scanner in order to show changes in brain activity involved in performing those tasks. Subjects are shown pictures of feet and other body parts, are asked to move their feet, and receive tactile (touch) stimulation of the foot or other body parts.

Control Subjects

One group of control subjects undergoes a single fMRI procedure. A second group of control subjects undergoes the same sequence of three fMRIs over the same time period as the amputee subjects. None of the control subjects undergo mirror therapy.

...

DETAILED DESCRIPTION:
Objective: The aim of this study is to investigate phantom limb pain (PLP), cortical reorganization and the modulation of PLP by visual input. Mirror therapy (viewing the intact limb in a mirror so that it appears to be the missing limb) has been shown to reduce PLP. This reduction demonstrates that vision can play a key role in modulating PLP. The study proposed here will identify brain regions critical for the success of this therapy using functional magnetic resonance imaging (fMRI).

Study population: Individuals with unilateral amputation of individual limbs and at least three episodes of PLP a week. Additionally, we will study amputees without PLP and healthy control volunteer subjects with no limb amputations.

Design: Amputee subjects with PLP will be scanned using fMRI while they undergo mirror therapy for PLP. During fMRI scans subjects will see images of hands or feet, move their limbs or experience tactile stimulation. Mirror therapy requires four weeks to be effective. Amputee subjects will be scanned prior to starting therapy, two weeks after starting mirror therapy and again after four weeks of mirror therapy. Mirror therapy sessions will be conducted daily and subjects will also complete daily questionnaires (Visual Analogue Scale, or VAS, and Short-Form McGill Pain Questionnaire or SF-MPQ) assessing their level of pain and number of PLP episodes. Amputees without PLP and one group of healthy control subjects will go through the same series of functional imaging scans over the same time period as the amputee subjects, allowing us to identify brain changes that may be associated with repeated scanning (e.g. due to practice of tasks) rather than resulting from the mirror therapy. Another group of control subjects will be scanned once to identify particular brain regions that might be involved in the integration of visual, motor and somatosensory information for use in the analysis of the amputee subject data.

Outcome measures: Changes in fMRI activation during the course of mirror therapy will be compared with data on the number of episodes of PLP, the average length of episodes, and the average intensity of pain assessed using the VAS and SF-MPQ. Analyses will focus on cortical regions known to be involved in visual, tactile and motor representations (including primary motor cortex, primary and secondary somatosensory cortex and regions of visual cortex selectively responsive during the viewing of body parts). Additional brain regions that might be involved in integrating visual, motor and somatosensory information will be identified in control subjects. Direct comparisons will be made between cortical regions (e.g. somatosensory regions) involved in the representation of the amputated limb compared with the intact limb and between amputee subject data and control subject data.

ELIGIBILITY:
* INCLUSION CRITERIA:

For amputee subjects with PLP:

* Male or female subjects, 18 to 75 years of age
* Written informed consent and written authorization for use or release of health and research study information
* Unilateral limb amputation
* Any level of prosthetic experience
* No prior history of vertebral disk disease/condition, sciatica or radiculopathy.
* No evidence of traumatic brain injury (TBI - permanent or temporary impairments of cognitive, physical and psychosocial functions with an associated diminished or altered state of consciousness)
* No known neurological disease or brain damage
* No neurological condition that would interfere with participation in the study
* Minimum of 3 phantom limb pain episodes each week
* Degree of pain evaluated by VAS scoring a minimum of 3 cm at time of screening for entry into study
* Ability to follow study instructions and likely to complete all required visits.

For amputee subjects without PLP:

* Male or female subjects, 18 to 75 years of age
* Written informed consent and written authorization for use or release of health and research study information
* Unilateral limb amputation
* Any level of prosthetic experience
* No prior history of vertebral disk disease/condition, sciatica or radiculopathy.
* No evidence of traumatic brain injury (TBI - permanent or temporary impairments of cognitive, physical and psychosocial functions with an associated diminished or altered state of consciousness)
* No known neurological disease or brain damage
* No neurological condition that would interfere with participation in the study
* No recurring episodes of PLP
* Ability to follow study instructions and likely to complete all required visits.

For healthy control subjects:

* Male or female subjects, 18 to 75 years of age.
* Written informed consent and written authorization for use or release of health and research study information.
* No prior history of vertebral disk disease/condition, sciatica or radiculopathy.
* Normal neurological examination.
* Ability to follow study instructions and likely to complete all required visits.

EXCLUSION CRITERIA:

For amputee subjects with PLP:

* Age less than 18 or greater than 75 years.
* Multiple limb amputation
* Amputation due to diabetes or vascular claudication
* Pending revision surgeries.
* Presence of embedded metallic shrapnel or other metal not compatible with MRIscanning.
* Presence of traumatic brain injury
* Known uncontrolled systemic disease- known cancer not in remission, known on-going infection, lupus, kidney disease requiring dialysis, any other systemic disease which might affect ability to participate in this study to its conclusion
* Concurrent participation in another investigational drug or device study for phantom limb pain or participation in the 30 days immediately prior to study enrollment.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Current Axis I or II diagnosis determined by a neurologist or psychiatrist in the 6 months prior to entry into the study.
* Subjects with lack of effort as determined by the neurologist or physiatrist. Subjects will be screened for effort using the Test of Memory Malingering (TOMM) first in order to exclude those with blatant exaggeration or malingering.
* Positive pregnancy test at the time of scanning (within 24 hours prior to the scheduled MRI scan, female subjects of child-bearing age will be given a pregnancy test)

For amputee subjects without PLP:

* Age less than 18 or greater than 75 years.
* Multiple limb amputation.
* Amputation due to diabetes or vascular claudication
* Pending revision surgeries.
* Presence of embedded metallic shrapnel or other metal not compatible with MRI scanning.
* Presence of traumatic brain injury
* Known uncontrolled systemic disease- known cancer not in remission, known on-going infection, lupus, kidney disease requiring dialysis, any other systemic disease which might affect ability to participate in this study to its conclusion
* Concurrent participation in another investigational drug or device study for phantom limb pain or participation in the 30 days immediately prior to study enrollment.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Current Axis I or II diagnosis determined by a neurologist or psychiatrist in the 6 months prior to entry into the study.
* Subjects with lack of effort as determined by the neurologist or physiatrist. Subjects will be screened for effort using the Test of Memory Malingering (TOMM) first in order to exclude those with blatant exaggeration or malingering.
* Positive pregnancy test at the time of scanning (within 24 hours prior to the scheduled MRI scan, female subjects of child-bearing age will be given a pregnancy test)

For healthy control subjects:

* Age less than 18 or greater than 75 years
* Presence of an amputation
* Presence of embedded metallic shrapnel or other metal not compatible with MRI scanning.
* Presence of traumatic brain injury
* Known uncontrolled systemic disease- known cancer not in remission, known on-going infection, lupus, kidney disease requiring dialysis, any other systemic disease which might affect ability to participate in this study to its conclusion
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study
* Current Axis I or II diagnosis determined by a neurologist or psychiatrist in the 6 months prior to entry into the study
* Positive pregnancy test at the time of scanning (within 24 hours prior to the scheduled MRI scan, female subjects of child-bearing age will be given a pregnancy test)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-03-05; Study Completion 2019-12-10

PRIMARY OUTCOMES:
Changes in fMRI signal

SECONDARY OUTCOMES:
Changes in pain measures

CONTACTS AND LOCATIONS:
Overall Officials: Christopher I Baker, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Ramachandran VS, Hirstein W. The perception of phantom limbs. The D. O. Hebb lecture. Brain. 1998 Sep;121 ( Pt 9):1603-30. doi: 10.1093/brain/121.9.1603. PMID 9762952
- [Background] Sherman RA, Sherman CJ, Parker L. Chronic phantom and stump pain among American veterans: results of a survey. Pain. 1984 Jan;18(1):83-95. doi: 10.1016/0304-3959(84)90128-3. PMID 6709380
- [Background] Jensen TS, Krebs B, Nielsen J, Rasmussen P. Phantom limb, phantom pain and stump pain in amputees during the first 6 months following limb amputation. Pain. 1983 Nov;17(3):243-256. doi: 10.1016/0304-3959(83)90097-0. PMID 6657285
- [Derived] Griffin SC, Curran S, Chan AWY, Finn SB, Baker CI, Pasquina PF, Tsao JW. Trajectory of phantom limb pain relief using mirror therapy: Retrospective analysis of two studies. Scand J Pain. 2017 Apr;15:98-103. doi: 10.1016/j.sjpain.2017.01.007. Epub 2017 Mar 7. PMID 28850360